CLINICAL TRIAL: NCT03054584
Title: Genetic Basis of Melanocytic Nevi
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 960347
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Melanocytic Nevi
MeSH Terms: conditions — Nevus, Pigmented

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collecting Nevi — Will be collecting Nevi and completing a DNA analysis, no intervention will be made.

SUMMARY:
The objective of this protocol is to further elucidate the genetic mutations that drive melanocytic nevi (benign melanocytic neoplasms, moles). This will be performed by whole genome, whole exome, or targeted sequencing of de-identified specimens.

Herein, the investigators plan to isolate DNA from de-identified skin biopsy specimens and blood samples:

1. From melanocytic nevi collected by skin biopsy (a shave or punch biopsy). A part of the tissue will be submitted for routine diagnostic dermatopathology and investigational histomorphologic and immunohistochemical analysis.
2. From corresponding normal tissue (blood). DNA isolated from blood will be used as a normal control when analyzing sequencing data to identify somatic mutations in lesional tissue.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects that are 18 years or older
* Subjects with melanocytic nevi\

Exclusion criteria:

* Patients less than 18 years of age
* Patients without melanocytic nevi
* Patients with a bleeding disorder or are taking anticoagulation medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seen in UC Davis dermatology clinic diagnosed as having melanocytic nevi will be recruited from the clinic during their routine visit. Subjects identified in clinic will be approached after their clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Genome Wide Mutation Analysis | Feb 2017 - December 2018
  Will be performing genome wide mutation analysis to quantify the number of mutations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No